CLINICAL TRIAL: NCT01417728
Title: Endomicroscopy for Assessment of Structural and Functional Changes in IBD Patients Treated With Anti-TNFalpha - Insights in the Process in Mucosal Healing
Brief Title: Endomicroscopy in IBD Patients
Acronym: EARLY
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Mudter2011
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: endomicroscopy; inflammatory bowel disease; mucosal healing; infliximab
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to analyze the mechanism of action of infliximab at the endomicroscopic level and to analyze mucosal healing - i.e. structural and functional changes in the mucosa in IBD patients - and associated processes such as permeability and bacterial invasion of the mucosa. In this study the role of the above mentioned parameters and further the establishment of endomicroscopic scores will serve to define new prognostic markers in view of long term remission upon infliximab treatment.

DETAILED DESCRIPTION:
The main goal of treatment for Crohn's disease and ulcerative colitis has always been the induction and maintenance of symptomatic improvement or at best remission. There is recent evidence that with immunosuppression and treatment with infliximab a long-term healing of the bowel can be achieved and that this affects the clinical outcome of both Crohn's disease and ulcerative colitis. Chronic idiopathic inflammatory bowel diseases (IBDs) including Crohn's disease, ulcerative colitis and indeterminate colitis are characterised by the presence of extensive areas of ulceration and inflammation in the gut. These ulcerations are the origin of several complications e.g fistulas, toxic megacolon, perforation and bleeding or developing neoplasias.

Therefore effective treatment of IBD should imply thoroughly and, if possible, complete healing of bowel ulcerations in parallel with clinical remission. There is evidence that infliximab, an immunoglobulin G1 monoclonal antibody against tumour necrosis factor, not only rapidly improves symptoms in patients with refractory IBDs, but also induces mucosal healing of ileocolonic lesions by week 4 after intravenous administration. The key question of course is whether healing of the mucosa of the bowel improves also the microstructural level of the mucosa and submucosa and perhaps translocation of commensal bacteria and barrier function as well. The validity of healing and maintain microscopic healing of the bowel mucosa and submucosa still has to be shown. Clinical studies showed that infliximab heals the mucosa of the colon in up to 60% by 8 weeks and maintains this healing for al long period of time. Unfortunately treatments that heal the mucosa do not cure Crohn's disease or ulcerative colitis; however, they are associated with a prolongation of the symptom free interval in comparison with the non-healed bowel. This fact suggests that the disease mechanism in the mucosa does not disappear with macroscopic healing of the ulcers and that the intraluminal trigger ends up damaging the mucosa again. For the purpose of clinical trials mucosal healing was defined so far by macroscopic view on the mucosa during white light endoscopy.

A microscopic analysis of the microstructure for assessment of healing seems to be necessary, especially to define objective end points for infliximab therapy to prevent relapses and complications. It is known that mucosal healing does not always correlate with clinical remission, therefore a microscopic diagnosis of ongoing inflammation is necessary.

Recently, a miniaturized confocal microscope was developed which could be integrated in the distal tip of a conventional colonoscope. This new diagnostic technology for gastrointestinal endoscopy, denoted confocal endomicroscopy, allowed in vivo histology of the mucosal layer during ongoing colonoscopy. Furthermore, in patients screened for sporadic colorectal cancer, surface and subsurface analysis at cellular and subcellular resolution could be used to predict intraepithelial neoplasias (INs) with high accuracy. Endomicroscopic image acquisition is performed by placing the tip of the colonoscope in direct contact with the targeted tissue site and providing in this manner surface and subsurface imaging at the time of ongoing video colonoscopy. It allows the detailed analysis of colorectal crypt architecture, deep vascular net structure and detailed mucosal / submucosal analysis. Studies in patients with ulcerative colitis showed that this novel endoscopic approach allowed to diagnose flat intraepithelial neoplasias with a high degree of accuracy and thus emerges as a crucial innovative imaging technology in the colon. Here, we propose to analyze the mucosa of patients with Crohn´s disease and ulcerative colitis before and after infliximab therapy using endomicroscopy for analysing microscopic healing processes during ongoing endoscopy.

ELIGIBILITY:
Inclusion criteria:

* Indication for therapy with infliximab according to the current guidelines.

Exclusion criteria:

* Inability to provide written informed consent
* Pregnancy or breast-feeding
* Severe uncontrolled coagulopathy
* Impaired renal function
* Known allergy to fluorescein

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: trusted IBD diagnosis (Crohn's disease of ulcerative colitis)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Assessment of mucosal healing changes by confocal laser endomicroscopy | 1 year
  Endomicroscopy will be used to assess the mucosal structure before and after treatment.
  Further Parameters:
  * assessment of mucosal barrier function in vivo during ongoing endoscopy
  * epithelial cell structure (development of new tools to differentiate mucosal structures and cells), e.g. crypt distortion, crypt lumen
  * infiltration of mononuclear cells
  * translocation of bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine I, University of Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Derived] Hundorfean G, Chiriac MT, Mihai S, Hartmann A, Mudter J, Neurath MF. Development and Validation of a Confocal Laser Endomicroscopy-Based Score for In Vivo Assessment of Mucosal Healing in Ulcerative Colitis Patients. Inflamm Bowel Dis. 2017 Dec 19;24(1):35-44. doi: 10.1093/ibd/izx012. PMID 29272480